CLINICAL TRIAL: NCT00483223
Title: A Phase II Study of Cisplatin or Carboplatin for Triple-Negative Metastatic Breast Cancer and Evaluation of p63/p73 as a Biomarker of Response
Brief Title: Platinum for Triple-Negative Metastatic Breast Cancer and Evaluation of p63/p73 as a Biomarker of Response
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other); Dana-Farber Cancer Institute (Other); North Shore Medical Center (Other)
Responsible Party: Principal Investigator, Steven Isakoff, MD, PhD, Attending Physician, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-412; TBCRC009 (Other: Translational Breast Cancer Research Consortium)
Record Dates: First submitted 2007-06-05; First posted 2007-06-06 (Estimated); Results first posted 2017-06-01 (Actual); Last update posted 2017-08-25 (Actual); Status verified 2017-07

CONDITIONS: Breast Cancer
Keywords: ER negative; PgR negative; HER2 negative; cisplatin; carboplatinum; platinum; p63; p73
MeSH Terms: conditions — Breast Neoplasms; Ectrodactyly, Ectodermal Dysplasia, and Cleft Lip-Palate Syndrome 3 | interventions — Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm (Experimental): Cisplatin or carboplatin (1 arm, 2 cohorts)
  Interventions: Drug: Cisplatin; Drug: carboplatin

INTERVENTIONS:
Drug: Cisplatin — Given intravenously on the first day of each 3-week treatment cycle at 75mg/m2. Participants may continue to receive study treatment as long as their disease does not worsen and they do not experience serious side effects.
  Other Names: Platinol
Drug: carboplatin — Given intravenously on the first day of each 3-week treatment cycle at AUC 6. Participants may continue to receive study treatment as long as their disease does not worsen and they do not experience serious side effects.
  Other Names: Paraplatin

SUMMARY:
The purpose of this research study is to :

* Determine how effective cisplatin or carboplatin is in slowing the time it takes for ER negative (estrogen-receptor-negative), PR negative (progesterone receptor-negative), HER2 negative (human epidermal growth factor receptor 2) breast cancer to progress. Cisplatin and carboplatin are anti-cancer chemotherapy drugs that stop cancer cells from growing abnormally and is used to treat other cancers.
* Evaluate a new biomarker to help determine which breast cancers are most likely to respond to cisplatin chemotherapy

The hypothesis is that Triple Negative metastatic breast cancer may be particularly sensitive to platinum, and that a subgroup of those patients may have a marker in their tumors that predicts response.

DETAILED DESCRIPTION:
This study is a Phase 2 study designed to evaluate cisplatin/carboplatin as first or second line therapy in metastatic triple negative (ER negative, PR negative, Her2 Negative) breast cancer and to evaluate the expression of p63/p73 as a biomarker to predict response.

* Participants will be given a cisplatin or carboplatin infusion intravenously on the first day of each treatment cycle. Each treatment cycle will last 3 weeks. Treating physician will select agent up to 41 patients in each cohort. Final primary endpoint analysis will use combined cis/carbo results.
* During all treatment cycles participants will have a physical exam (including weight and vital signs) and they will be asked general questions about their health and any medications they may be taking, as well as specific questions about any side effects they may be experiencing while receiving study treatment.
* During every treatment cycle participants will have standard blood tests to check blood counts, liver and kidney function, and a blood marker for you particular type of cancer.
* CT scans will be taken of the participants tumor every 2 to 3 cycles to assess the response of the tumor to cisplatin.
* Participants will be in this study for as long as they tolerate the study treatment and their disease does not get any worse.
* Participants will be required to have a sample of their original tumor sent to Massachusetts General Hospital for correlative studies, or a sample from a metastatic diagnostic biopsy.
* Patients with accessible tumor will be asked to provide an optional metastatic tumor biopsy for correlative studies.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive breast cancer with stage IV disease, according to AJCC 6th edition (American Joint Committee on Cancer), either biopsy proven or with unequivocal evidence of metastatic disease by physical examination or radiological study
* All tumors must be ER-, PGR- and HER2-negative
* 18 years of age or older
* Paraffin tissue block is required from the primary tumor tissue or from diagnostic metastatic biopsy at time of relapse
* Measurable disease by RECIST
* Performance status of 0,1 or 2 by ECOG criteria (Eastern Cooperative Oncology Group)
* Life expectancy greater than 12 weeks
* Normal organ and bone marrow function documented within 14 days prior to enrollment as defined by the protocol

Exclusion Criteria:

* More than 1 prior chemotherapy for the treatment of recurrent or metastatic breast cancer
* Prior treatment with cisplatin, carboplatin, or other platinum chemotherapy agents
* Active brain metastases or unevaluated neurological symptoms suggestive of brain metastases
* Intercurrent illness or other major medical condition or comorbid condition that might affect study participation
* Significant history of uncontrolled cardiac disease such as uncontrolled hypertension, unstable angina, recent myocardial infarction, uncontrolled congestive heart failure, cardiomyopathy either symptomatic or asymptomatic but with decreased ejection fraction <45%
* Renal dysfunction for which cisplatin dose would either require dose modification or would be considered unsafe
* Pregnant or nursing women
* History or other malignancy that was not treated with curative intent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2007-06; Primary Completion 2014-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Isakoff, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (10):
- United States (10):
  - University of Alabama-Birmingham, Birmingham, Alabama
  - UCSF, San Francisco, California
  - Georgetown - Lombardi Cancer Center, Washington D.C., District of Columbia
  - Johns Hopkins University Medical Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - North Shore Medical Center, Peabody, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Isakoff SJ, Mayer EL, He L, Traina TA, Carey LA, Krag KJ, Rugo HS, Liu MC, Stearns V, Come SE, Timms KM, Hartman AR, Borger DR, Finkelstein DM, Garber JE, Ryan PD, Winer EP, Goss PE, Ellisen LW. TBCRC009: A Multicenter Phase II Clinical Trial of Platinum Monotherapy With Biomarker Assessment in Metastatic Triple-Negative Breast Cancer. J Clin Oncol. 2015 Jun 10;33(17):1902-9. doi: 10.1200/JCO.2014.57.6660. Epub 2015 Apr 6. PMID 25847936

RESULTS

PARTICIPANT FLOW:
Groups:
- Cisplatin or Carboplatin: Cisplatin or carboplatin (1 arm, 2 cohorts)
  Cisplatin: Given intravenously on the first day of each 3-week treatment cycle at 75mg/m2. Participants may continue to receive study treatment as long as their disease does not worsen and they do not experience serious side effects.
  carboplatin: Given intravenously on the first day of each 3-week treatment cycle at AUC 6. Participants may continue to receive study treatment as long as their disease does not worsen and they do not experience serious side effects.
Period: Overall Study
Arm/Group | Cisplatin or Carboplatin
Started | 86
Completed | 86
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm
Number analyzed (Participants) | 86
Age, Continuous [Median (Full Range); unit: years] | 52 [30 to 78]
Age, Customized [Count of Participants; unit: Participants]
  < 40 | 13
  40-65 | 63
  > 65 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 69
  African American | 7
  Asian | 4
  > one or other | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 86
ECOG PS [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group performance score. The performance scale describes a participants level of functioning in terms of their ability to care for themselves. daily activity, and physical ability.
  0. Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  Participants
    0 | 55
    1 | 20
    2 | 5
    Not reported | 6
Site of metastases [Number; unit: participants] — The number of participants with metastases at the specified cites.
  participants
    Lymph nodes | 54
    Lung | 44
    Bone | 25
    Liver | 25
    Skin | 16
    Brain | 4
Stage at initial diagnosis of breast cancer [Count of Participants; unit: Participants] — This describes the stage of breast cancer at diagnosis according to the American Joint Commission on Cancer (AJCC) Version 7. Generally, stage 1 is a cancer that is less than 2 cm and lymph node negative, stage 2 is a tumor between 2-5 cm and/or 1-3 lymph nodes positive, and stage 3 is a tumor with more than 3 lymph nodes positive or a tumor invading the skin. Stage 4 indicates that the cancer has spread into distant parts of the body. In general, lower stage cancers have a better prognosis, and higher stage cancers are more advanced.
  Participants
    1 | 10
    2 | 32
    3 | 37
    4 | 7
Prior chemotherapy [Number; unit: participants] — The prior chemotherapy received by the participants.The rows represent the number of participants that received any adjuvant/neoadjuvant as well as the number of participant that received Anthracycline or Taxane as their adjuvant/neoadjuvant drug.
  participants
    Adjuvant/neoadjuvant | 74
    Anthracycline | 65
    Taxane | 67
Treatment cohort [Count of Participants; unit: Participants] — The number of participants assigned to each treatment cohort within the single arm of this study.
  Participants
    Cisplatin (cohort 1) | 43
    Carboplatin (cohort 2) | 43

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Objective response rate (ORR) (complete response [CR]+ partial response [PR]) by RECIST (Response Evaluation Criteria In Solid Tumors).
  Complete Response (CR): Disappearance of all target lesions
  Partial Response (PR): At least a 30% decrease in the sum of the LD (longest diameter) of target lesions, taking as reference the baseline sum LD
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started
  Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cisplatin or Carboplatin
Number analyzed (Participants) | 86
Participants
  Complete Response | 3
  Partial Response | 19
  Stable Disease > 6 Months | 4
  Progressive Disease | 57
  Not Evaluable | 3

2. Primary Outcome: Response Rate Categorized by p63/p73 Ratio
Description: Response rate categorized by pre-specified ΔNp63/TAp73 expression ratio cutoff in the primary tumors from this patient cohort as a bio-marker to predict response to cisplatin or carboplatin. Response is defined as partial or completed response as determined by RECIST. Expression ratio was measured using quantitative RT-PCR (Reverse transcription polymerase chain reaction).
Time Frame: 3 years
Population: Patients from either cohort with a tumor sample available to evaluate for expression ratio.
Measure: Count of Participants; unit: Participants
Arm/Group | Cisplatin or Carboplatin
Number analyzed (Participants) | 61
Participants
  p63/p73 > 2: number analyzed (Participants) | 33
  p63/p73 > 2: Response | 9
  p63/p73 > 2: No Response | 24
  p63/p73 < 2: number analyzed (Participants) | 28
  p63/p73 < 2: Response | 5
  p63/p73 < 2: No Response | 23
Statistical Analysis 1: Comparison: Cisplatin or Carboplatin; H0: no association between expression ratio and response rate Ha: Participants with expression ratio greater than 2 would have higher response rate; Test type: Other; p = 0.54, t-test, 2 sided

3. Secondary Outcome: Objective Response Rate Categorized by Subgroup
Description: The number of participants achieving an objective response (as determined by RECIST) categorized by treatment cohort and whether the treatment was first or second line treatment. First line treatment means that the drug used was the first drug used for the treatment of the primary cancer. Second line treatment means that a first line treatment failed to produce the desired response, so a new drug was used for treatment.
Time Frame: 3 years
Population: Response rate is divide by drug cohort and categorized by first or second-line treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Cisplatin or Carboplatin
Number analyzed (Participants) | 86
Participants
  Cisplatin: number analyzed (Participants) | 43
  Cisplatin: First line: Response | 12
  Cisplatin: First line: No response | 22
  Cisplatin: Second line: Response | 2
  Cisplatin: Second line: No response | 7
  Carboplatin: number analyzed (Participants) | 43
  Carboplatin: First line: Response | 8
  Carboplatin: First line: No response | 27
  Carboplatin: Second line: Response | 0
  Carboplatin: Second line: No response | 8

4. Secondary Outcome: Progression Free Survival and Overall Survival
Description: Median progression free survival and overall survival (progression determined using RECIST) during a median follow-up time of 50 months.
Time Frame: 5 years
Measure: Median (Full Range); unit: Months
Arm/Group | Cisplatin or Carboplatin
Number analyzed (Participants) | 86
Months
  Median Progression Free Survival | 2.9 [0.1 to 56.8]
  Median Overall Survival | 11 [1.6 to 56.8]

ADVERSE EVENTS:
Time Frame: On day 1 of each 21 day treatment cycle for duration of treatment.
Description: Physical exam, laboratory test, and questions are used to assess adverse events on the first day of every 21 day cycle.
Arm/Group | Cisplatin or Carboplatin
All-Cause Mortality (participants affected / at risk) | 75/86
Serious Adverse Events (participants affected / at risk) | 8/86
Other Adverse Events (participants affected / at risk) | 85/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cisplatin or Carboplatin (N=86)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Neutrophil Count (Investigations) | 1 (1)
Infection with normal ANC (Infections and infestations) | 4 (4)
Hypersensitivity reaction to Cisplatin (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cisplatin or Carboplatin (N=86)
Allergic reaction (Immune system disorders) | 4 (7)
Tinnitus (Ear and labyrinth disorders) | 16 (34)
Hemoglobin (Investigations) | 63 (250)
Leukocytes (Investigations) | 34 (97)
Lymphopenia (Investigations) | 20 (71)
Neutrophils (Investigations) | 35 (75)
Platelets (Investigations) | 28 (72)
Fatigue (General disorders) | 57 (217)
Fever w/o neutropenia (General disorders) | 8 (8)
Insomnia (Psychiatric disorders) | 10 (35)
Constitutional, other (General disorders) | 7 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (12)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 4 (10)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 9 (17)
Hot flashes (Vascular disorders) | 8 (25)
Anorexia (Metabolism and nutrition disorders) | 15 (22)
Constipation (Gastrointestinal disorders) | 26 (61)
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 9 (13)
Nausea (Gastrointestinal disorders) | 57 (143)
Vomiting (Gastrointestinal disorders) | 16 (29)
GI-other (Gastrointestinal disorders) | 6 (9)
Febrile neutropenia (Blood and lymphatic system disorders) | 11 (21)
Edema limb (General disorders) | 10 (19)
Hypoalbuminemia (Metabolism and nutrition disorders) | 10 (14)
Alkaline phosphatase (Metabolism and nutrition disorders) | 19 (51)
ALT, SGPT (Metabolism and nutrition disorders) | 16 (28)
AST, SGOT (Metabolism and nutrition disorders) | 25 (51)
Hypocalcemia (Metabolism and nutrition disorders) | 12 (14)
Hyperglycemia (Metabolism and nutrition disorders) | 39 (79)
Hypomagnesemia (Metabolism and nutrition disorders) | 28 (105)
Hypokalemia (Metabolism and nutrition disorders) | 9 (19)
Hyponatremia (Metabolism and nutrition disorders) | 15 (27)
Dizziness (Nervous system disorders) | 10 (14)
Anxiety (Psychiatric disorders) | 8 (19)
Depression (Psychiatric disorders) | 4 (7)
Neuropathy-sensory (Nervous system disorders) | 32 (114)
Neuropathy-peripheral (Nervous system disorders) | 5 (10)
Neurologic-other (Nervous system disorders) | 5 (8)
Abdomen, pain (Gastrointestinal disorders) | 9 (11)
Back, pain (Musculoskeletal and connective tissue disorders) | 11 (20)
Bone, pain (Musculoskeletal and connective tissue disorders) | 6 (10)
Chest wall, pain (Musculoskeletal and connective tissue disorders) | 10 (11)
Chest/thoracic pain NOS (Musculoskeletal and connective tissue disorders) | 4 (8)
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 6 (12)
Head/headache (Nervous system disorders) | 12 (21)
Joint, pain (Musculoskeletal and connective tissue disorders) | 7 (9)
Muscle, pain (Musculoskeletal and connective tissue disorders) | 5 (10)
Neck, pain (Musculoskeletal and connective tissue disorders) | 5 (6)
Pain-other (General disorders) | 9 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (25)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 25 (52)
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes